CLINICAL TRIAL: NCT03256019
Title: Improvement of Recovery of Spontaneous Circulation and Survival Using the Video-laryngoscopy for out-of Hospital Cardiac Arrest Patient
Brief Title: Compare Outcomes of CPR Between the Video-laryngoscopy (VL) Users and the Direct-laryngoscopy (DL) Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Sang O, Park, Associate Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPRIntuVLvsDL
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Cardiopulmonary Arrest
Keywords: intubation; Cardiopulmonary Resuscitation
MeSH Terms: conditions — Heart Arrest | interventions — Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DL user (Active Comparator): Experienced emergency physicians who primarily used the direct laryngoscopy (DL) for endotracheal intubation during cardiopulmonary resuscitation.
  Interventions: Procedure: Endotracheal Intubation
- VL user (Active Comparator): Experienced emergency physicians who primarily used the videolaryngoscopy (VL) for endotracheal intubation during cardiopulmonary resuscitation.
  Interventions: Procedure: Endotracheal Intubation

INTERVENTIONS:
Procedure: Endotracheal Intubation — Insertion of endotracheal tube into the trachea and supply oxygen using the Ambu-bagging during cardiopulmonary resuscitation

SUMMARY:
This is a clinical study based on the analysis of video-clip data of cardiopulmonary resuscitation (CPR) and clinical data for out of hospital cardiac arrest patients between 2011 and 2015. Aim of study is to compare the endotracheal intubation performance and CPR outcomes between videolaryngoscopy (VL) and direct laryngoscopy (DL) users.

DETAILED DESCRIPTION:
Endotracheal intubation (ETI) has been considered to be the best method of airway management during cardiopulmonary resuscitation (CPR). However ETI during CPR is a highly skill-dependent procedure, then it should be attempted only highly trained physicians. Because of technical difficulty in using direct laryngoscopy (DL), various types of videolaryngoscopy (VL) devices using micro-camera technology have been designed to overcome the problems of DL.

This study tried to compare the recovery of spontaneous circulation (ROSC) and survival discharge between use of standard device (DL) and VL in a real clinical setting. In addition, this study also compare the first pass success rate of ETI,speed of ETI, incidences of complications, and chest compression interruptions during cardiopulmonary resuscitation between both device users.

ELIGIBILITY:
Inclusion Criteria:

* Patients who suffer sudden out-of hospital cardiac arrest

Exclusion Criteria:

* Cardiac arrests from multiple trauma
* Cases of requesting the do-not attempt resuscitation before ETI
* Intubated cases before arrival to emergency department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Survival with good neurologic outcome | 6 months after emergency department visit
  Survived patients who were conscious and able to perform independent activities of daily life (CPC1 or CPC2)

SECONDARY OUTCOMES:
ROSC | within 1 hour after emergency department visit
  Recovery of spontaneous circulation by successful resuscitation
total time to complete ETI from the beginning | within 1 hour after emergency department visit
  time from the advancement of the blade into the patient's mouth to the delivery of the first successful ventilation using the bag
complication | within 1 hour after emergency department visit
  Presence of chest compression interruption, esophageal intubation and dental injuries

CONTACTS AND LOCATIONS:
Overall Officials: Sang O Park, M.D,Ph.D, Principal Investigator — Department of Emergency Medicine, Konkuk University Medical center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soar J, Nolan JP, Bottiger BW, Perkins GD, Lott C, Carli P, Pellis T, Sandroni C, Skrifvars MB, Smith GB, Sunde K, Deakin CD; Adult advanced life support section Collaborators. European Resuscitation Council Guidelines for Resuscitation 2015: Section 3. Adult advanced life support. Resuscitation. 2015 Oct;95:100-47. doi: 10.1016/j.resuscitation.2015.07.016. No abstract available. PMID 26477701
- [Background] Hasegawa K, Hiraide A, Chang Y, Brown DF. Association of prehospital advanced airway management with neurologic outcome and survival in patients with out-of-hospital cardiac arrest. JAMA. 2013 Jan 16;309(3):257-66. doi: 10.1001/jama.2012.187612. PMID 23321764
- [Background] Wang HE, Simeone SJ, Weaver MD, Callaway CW. Interruptions in cardiopulmonary resuscitation from paramedic endotracheal intubation. Ann Emerg Med. 2009 Nov;54(5):645-652.e1. doi: 10.1016/j.annemergmed.2009.05.024. Epub 2009 Jul 2. PMID 19573949
- [Background] Kaplan MB, Ward DS, Berci G. A new video laryngoscope-an aid to intubation and teaching. J Clin Anesth. 2002 Dec;14(8):620-6. doi: 10.1016/s0952-8180(02)00457-9. PMID 12565125
- [Background] Rothfield KP, Russo SG. Videolaryngoscopy: should it replace direct laryngoscopy? a pro-con debate. J Clin Anesth. 2012 Nov;24(7):593-7. doi: 10.1016/j.jclinane.2012.04.005. PMID 23101777